CLINICAL TRIAL: NCT02724020
Title: A Phase 2, Open-label Study to Evaluate the Efficacy and Safety of Single-Agent MLN0128 and the Combination of MLN0128+MLN1117 Compared With Everolimus in the Treatment of Adult Patients With Advanced or Metastatic Clear-Cell Renal Cell Carcinoma That Has Progressed on Vascular Endothelial Growth Factor-Targeted Therapy
Brief Title: MLN0128 and MLN0128 + MLN1117 Compared With Everolimus in the Treatment of Adults With Advanced or Metastatic Clear-Cell Renal Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C31005; 2015-002133-22 (EudraCT Number); U1111-1172-1808 (Registry Identifier: WHO)
Record Dates: First submitted 2016-03-25; First posted 2016-03-31 (Estimated); Results first posted 2021-02-21 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Clear-cell Metastatic Renal Cell Carcinoma
Keywords: Drug therapy
MeSH Terms: conditions — Clear-cell metastatic renal cell carcinoma | interventions — Everolimus; sapanisertib; serabelisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A: Single-agent Everolimus 10 mg QD (Active Comparator): Everolimus 10 mg capsules, orally, once daily in a 28-day treatment cycle until disease progression, consent withdrawal, death, or transfer to the Post-trial Access (PTA) program (Median duration of treatment was 15.43 weeks up to end of study).
  Interventions: Drug: Everolimus
- Arm B: Single-agent MLN0128 30 mg QW (Experimental): MLN0128 30 mg capsules, orally, once weekly on Days 1, 8, 15, and 22 of a 28-day treatment cycle until disease progression, unacceptable toxicity, consent withdrawal, death, or transfer to the PTA program (Median duration of treatment was 9.64 weeks up to end of study).
  Interventions: Drug: MLN0128
- Arm C: Combination of MLN0128 4 mg QD + MLN1117 200 mg QD (Experimental): MLN0128 4 mg and MLN1117 200 mg capsules, orally, both once daily for 3 days per week (QD X 3) on Days 1-3, 8-10, 15-17, and 22-24 of a 28-day treatment cycle until disease progression, unacceptable toxicity, consent withdrawal, death, or transfer to the PTA program (Median duration of treatment was 9.43 weeks up to end of study).
  Interventions: Drug: MLN0128; Drug: MLN1117

INTERVENTIONS:
Drug: Everolimus — Everolimus capsules.
  Arms: Arm A: Single-agent Everolimus 10 mg QD
Drug: MLN0128 — MLN0128 capsules.
  Other Names: TAK-228; INK0128
  Arms: Arm B: Single-agent MLN0128 30 mg QW; Arm C: Combination of MLN0128 4 mg QD + MLN1117 200 mg QD
Drug: MLN1117 — MLN1117 capsules.
  Other Names: TAK-117; INK1117
  Arms: Arm C: Combination of MLN0128 4 mg QD + MLN1117 200 mg QD

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of single-agent MLN0128 and the combination of MLN0128 + MLN1117 compared with everolimus in the treatment of participants with metastatic clear-cell renal cell carcinoma (mccRCC) that have progressed on vascular endothelial growth factor (VEGF)-targeted therapy.

DETAILED DESCRIPTION:
The drugs being tested in this study are called MLN0128 and MLN1117. MLN0128 and MLN1117 are being tested to treat people who have mccRCC. This study will assess the efficacy and safety of MLN0128 and MLN1117 as well as how it is processed by the body in participants with advanced or mccRCC.

The study will enroll approximately 96 participants. Participants will be randomly assigned (by chance, like flipping a coin) to one of the three treatment groups:

* Everolimus 10 mg once daily
* MLN0128 30 mg once weekly
* MLN0128 4 mg once daily for 3 days per week + MLN1117 200 mg once daily for 3 days per week

All participants will be asked to take the study drug at the same time on each scheduled day.

This multi-center trial will be conducted worldwide. The overall time to participate in this study is 2 years after last participant is randomized, or when the last participant discontinues study treatment (approximately 3 years). Participants will make multiple visits to the clinic including a follow-up visit 30 to 40 days after receiving their last dose of study drug or prior to start of subsequent anticancer therapy for safety assessment. Participants will then be followed for Progression Free and Overall Survival.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants aged 18 years or older.
2. Histologically confirmed renal cell carcinoma (RCC) with a clear-cell component.
3. Evidence that the RCC is advanced or metastatic.
4. Radiologic evidence of PD (according to RECIST Version 1.1) either during or within 6 months after stopping their most recent systemic therapy for RCC before enrollment into this study.
5. At least 1, prior line of VEGF-targeted therapy, but not more than 4 total prior lines of systemic therapy. Exposure to more than 1 line of VEGF-targeted therapy is acceptable. Participants may also have received prior therapies with interferon, interleukin 2 (IL-2), anti-PD1 antibodies, cabozantinib or other experimental agents, but not prior therapy with any agent that targets phosphoinositide 3-kinase (PI3K), serine/ threonine-specific protein kinase (AKT), or mechanistic (or mammalian) target of rapamycin (mTOR).
6. Karnofsky Performance Status (KPS) greater than or equal to (>=) 70%.
7. Life expectancy of >=3 months.
8. Female participants who:

   * Are postmenopausal for at least 1 year before the screening visit, OR
   * Are surgically sterile, OR
   * If they are of childbearing potential, agree to practice 1 highly effective method of contraception, and 1 additional effective (barrier) method, at the same time, from the time of signing the informed consent through 90 days (or longer, as mandated by local labelling [example, United States Prescribing Information (USPI), Summary of Product Characteristics (SmPC), etc;]) after the last dose of study drug, OR
   * Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the participant. (Periodic abstinence [example, calendar, ovulation, symptothermal, postovulation methods], withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception. Female and male condoms should not be used together.).

   Male participants, even if surgically sterilized (that is, status postvasectomy), who:
   * Agree to practice highly effective barrier contraception during the entire study treatment period and through 120 days after the last dose of study drug (or longer, as mandated by local labelling [example, USPI, SmPC, etc]), OR
   * Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the participant (Periodic abstinence [example, calendar, ovulation, symptothermal, postovulation methods for the female partner], withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception. Female and male condoms should not be used together.).
   * Agree not to donate sperm during the course of this study or within 120 days after receiving their last dose of study drug.
9. Suitable venous access for the study-required blood sampling.
10. Screening clinical laboratory values:

    * Absolute neutrophil count >=2000 per microliter (/mcL) and platelet count >=100,000/mcL;
    * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) less than or equal to (<=) 2.5*the upper limit of normal (ULN);
    * Total bilirubin <=1.5*ULN;
    * Estimated creatinine clearance by Cockcroft-Gault >=40 milliliter per minute (mL/min) / 1.73 square meter (m^2);
    * Glycosylated hemoglobin (HbA1c) less than (<) 7.0%, fasting serum glucose <=130 milligram per deciliter (mg/dL), and fasting triglycerides <=300 mg/dL.
11. At least 14 days since the end of prior systemic VEGF-targeted treatment (that is, sunitinib, pazopanib, axitinib, or sorafenib), radiotherapy, or surgical procedure with resolution of all treatment-related toxicity (except alopecia and hypothyroidism) either to Grade 0 or 1 (National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE] Version 4.03) or to baseline.
12. At least 21 days since the last dose of bevacizumab, other antibody, or interferon.
13. Voluntary written consent given before performance of any study-related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the participant at any time without prejudice to future medical care.

Exclusion Criteria:

1. Central nervous system (CNS) metastasis.
2. Other clinically significant co-morbidities, such as uncontrolled pulmonary disease, active CNS disease, active infection, or any other condition that might compromise the participant's participation in the study.
3. Known human immunodeficiency virus infection.
4. Known hepatitis B surface antigen-positive, or known or suspected active hepatitis C infection.
5. Manifestations of malabsorption due to prior gastrointestinal (GI) surgery, GI disease, or for an unknown reason that may alter the absorption of everolimus, MLN0128, or MLN1117. In addition, participants with enteric stomata are excluded.
6. Women who are either breast feeding or pregnant.
7. History of any of the following within the last 6 months before administration of the first dose of study drug

   * Ischemic myocardial event, including angina requiring therapy and artery revascularization procedures;
   * Ischemic cerebrovascular event, including transient ischemic attack and artery revascularization procedures;
   * Requirement for inotropic support (excluding digoxin), or serious (uncontrolled) cardiac arrhythmia (including atrial flutter/fibrillation, ventricular fibrillation, or ventricular tachycardia);
   * Placement of a pacemaker for control of rhythm;
   * New York Heart Association Class III or IV heart failure;
   * Pulmonary embolism.
8. Significant active cardiovascular or pulmonary disease including:

   * Uncontrolled hypertension (that is, either systolic blood pressure greater than [>] 160 millimeter of mercury [mm Hg]; diastolic blood pressure >95 mm Hg). Use of anti-hypertensive agents to control hypertension before Cycle 1 Day 1 is allowed;
   * Pulmonary hypertension.
   * Uncontrolled asthma or oxygen saturation <90% by arterial blood gas analysis or pulse oximetry on room air.
   * Significant valvular disease; severe regurgitation or stenosis by imaging independent of symptom control with medical intervention; or history of valve replacement.
   * Medically significant (symptomatic) bradycardia.
   * History of arrhythmia requiring an implantable cardiac defibrillator.
   * Baseline prolongation of the rate-corrected QT interval (QTc; example, repeated demonstration of QTc interval >480 millisecond [ms], or history of congenital, long-QT syndrome, or torsades de pointes).
9. Diagnosed or treated for another malignancy within 2 years before administration of the first dose of study drug, or previously diagnosed with another malignancy and have any evidence of residual disease. Participants with nonmelanoma skin cancer, superficial bladder cancer, very low risk prostate on observation, or carcinoma in situ of any type are not excluded if they have undergone complete resection.
10. Prior therapy with agents that target Phosphatidylinositide 3-kinases (PI3K), Protein kinase B (AKT), or mechanistic target of rapamycin (mTOR). Participants with known hypersensitivity to everolimus or rapamycin derivatives are also excluded.
11. Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol.
12. Participants who have taken a proton pump inhibitor (PPI) within 3 days before receiving the first dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2016-06-30 (Actual); Primary Completion 2020-02-03 (Actual); Study Completion 2020-10-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (36):
- United States (7):
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - Florida Cancer Specialists-Broadway, Venice, Florida
  - Florida Cancer Specialists, West Palm Beach, Florida
  - Hackensack University Medical Center PARTNER, Hackensack, New Jersey
  - The Ohio State University Comprehensive Cancer Center Arthur G. James Cancer Hospital, Columbus, Ohio
  - Tennessee Oncology, Nashville, Tennessee
  - The Center for Cancer and Blood Disorders, Weatherford, Texas
- Canada (2):
  - CancerCare Manitoba, Winnipeg, Manitoba
  - McMaster University, Hamilton, Ontario
- Czechia (3):
  - Fakultni nemocnice u sv. Anny v Brne, Brno
  - Fakultni nemocnice Olomouc, Olomouc
  - Fakultni nemocnice v Motole, Prague
- France (5):
  - Groupe Hospitalier Saint Andre - Hopital Saint Andre, Bordeaux, Aquitaine
  - ICL-Alexis Vautrin, Departement dOncologie Medicale, Vandœuvre-lès-Nancy, Meurthe Et Moselle
  - Groupe Hospitalier Pitie-Salpetriere, Paris, Paris
  - Institut de Cancerologie de l'Ouest Paul Papin, Angers, Pays de la Loire Region
  - Clinique Victor Hugo - Centre Jean Bernard, Le Mans, Sarthe
- Italy (4):
  - Azienda Ospedaliera Universitaria Policlinico Sant'Orsola Malpighi, Bologna
  - Istituto Nazionale Tumori Fondazione G. Pascale, Napoli
  - IOV - Istituto Oncologico Veneto IRCCS, Padua
  - Fondazione IRCCS Policlinico San Matteo, Pavia
- Poland (2):
  - Beskidzkie Centrum Onkologii im.Jana Pawla II, Bielsko-Biala
  - Instytut MSF, Ulica Pilota Stanislawa Wigury 19, Lodz
- Spain (7):
  - Hospital Duran i Reynals, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clinic i Provincial de Barcelona, Barcelona
  - MD Anderson Cancer Centre, Madrid
  - Hospital Universitario Ramon Y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
- United Kingdom (6):
  - Royal Devon and Exeter Hospital (Wonford), Exeter, Devon
  - Lancashire Teaching Hospitals NHS Foundation Trust, Blackburn, England
  - Barts Hospital, London, Greater London
  - The Christie, Manchester, Greater Manchester
  - Velindre Cancer Centre, Cardiff, South Glamorgan
  - Royal Surrey County Hospital, Guildford, Surrey

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at approximately 60-70 investigative sites in Czech Republic, France, Italy, Poland, Spain, United Kingdom, Canada and United States from 30 June 2016 to 13 October 2020.
Pre-assignment Details: Participants with a diagnosis of metastatic clear-cell renal cell carcinoma were randomized at a ratio of 1:1:1 to open label treatment period with single-agent MLN0128 and the combination of MLN0128 and MLN1117 compared with single-agent everolimus.
Period: Overall Study
Arm/Group | Arm A: Single-agent Everolimus 10 mg QD | Arm B: Single-agent MLN0128 30 mg QW | Arm C: Combination of MLN0128 4 mg QD + MLN1117 200 mg QD
Started | 32 | 32 | 32
Treated (Safety Analysis Set) | 32 | 32 | 31
Completed | 0 | 0 | 0
Not Completed | 32 | 32 | 32
Not completed — Death | 16 | 18 | 19
Not completed — Lost to Follow-up | 0 | 3 | 0
Not completed — Site Terminated by Sponsor | 15 | 8 | 8
Not completed — Withdrawal by Subject | 1 | 3 | 5

BASELINE CHARACTERISTICS:
Population: Full Analysis Set included all randomized participants.
Groups:
- Arm C: Combination of MLN0128 4 mg QD + MLN1117 200 mg QD: MLN0128 4 mg and MLN1117 200 mg capsules, orally, both once daily for 3 days per week (QD X 3) on Days 1-3, 8-10, 15-17, and 22-24 of a 28-day treatment cycle until disease progression, unacceptable toxicity, consent withdrawal, death, or transfer to the PTA (Median duration of treatment was 9.43 weeks up to end of study).
- Total: Total of all reporting groups
Arm/Group | Arm A: Single-agent Everolimus 10 mg QD | Arm B: Single-agent MLN0128 30 mg QW | Arm C: Combination of MLN0128 4 mg QD + MLN1117 200 mg QD | Total
Number analyzed (Participants) | 32 | 32 | 32 | 96
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.7 (11.41) | 61.6 (8.90) | 63.3 (9.06) | 63.2 (9.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 10 | 7 | 23
  Male | 26 | 22 | 25 | 73
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 2 | 2
  Not Hispanic or Latino | 28 | 30 | 27 | 85
  Unknown or Not Reported | 4 | 2 | 3 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1
  White | 27 | 29 | 27 | 83
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 4 | 3 | 4 | 11
Region of Enrollment [Count of Participants; unit: Participants]
  Czech Republic | 1 | 1 | 2 | 4
  France | 4 | 2 | 2 | 8
  Italy | 11 | 9 | 4 | 24
  Poland | 2 | 2 | 1 | 5
  Spain | 6 | 6 | 7 | 19
  United Kingdom | 4 | 4 | 9 | 17
  Canada | 2 | 1 | 2 | 5
  United States | 2 | 7 | 5 | 14
Height [Mean (Standard Deviation); unit: cm] — Population: Number analyzed is the number of participants with data available for height at Baseline.
  cm
    number analyzed (Participants) | 31 | 32 | 31 | 94
    (all) | 170.23 (8.489) | 171.16 (10.626) | 172.01 (8.349) | 171.13 (9.159)
Weight [Mean (Standard Deviation); unit: kg] — Population: Number analyzed is the number of participants with data available for weight at Baseline.
  kg
    number analyzed (Participants) | 31 | 32 | 32 | 95
    (all) | 75.69 (12.449) | 78.12 (15.473) | 80.40 (17.896) | 78.10 (15.419)

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as the time from the date of randomization to the date of first documentation of progressive disease (PD) or death due to any cause, whichever occurs first. Per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria. PD was defined as at least a 20% increase in the sum of the longest diameter (LD) of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: From first dose of study drug up to disease progression or death, assessed up to 43 months
Population: Full Analysis Set included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Single-agent Everolimus 10 mg QD | Arm B: Single-agent MLN0128 30 mg QW | Arm C: Combination of MLN0128 4 mg QD + MLN1117 200 mg QD
Number analyzed (Participants) | 32 | 32 | 32
months | 3.8 [2.0 to 5.4] | 3.6 [1.9 to 5.7] | 3.1 [1.9 to 5.4]
Statistical Analysis 1: Comparison: Arm A: Single-agent Everolimus 10 mg QD vs Arm B: Single-agent MLN0128 30 mg QW; Test type: Superiority; p = 0.388, Stratified Log-rank Test; Hazard Ratio (HR) = 1.33, 95% CI 2-sided [0.75 to 2.36] — HR obtained by stratified Cox proportion hazard model adjusted for prior lines of therapy and the international metastatic renal cell carcinoma database consortium risk category. A hazard ratio < 1 indicated an advantage compared to Everolimus
Statistical Analysis 2: Comparison: Arm A: Single-agent Everolimus 10 mg QD vs Arm C: Combination of MLN0128 4 mg QD + MLN1117 200 mg QD; Test type: Superiority; p = 0.667, Stratified Log-rank Test; Hazard Ratio (HR) = 1.37, 95% CI 2-sided [0.75 to 2.52] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An AE was defined as any untoward medical occurrence in participants administered a pharmaceutical product; the untoward medical occurrence does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product whether or not it is related to the medicinal product. TEAE was defined as the event that occur after administration of the first dose of study drug and through 30 days after the last dose of study drug.
Time Frame: From first dose of study drug through 30 days after the last dose of study drug (approximately up to 31 months)
Population: Safety Analysis Set included participants who receive at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Single-agent Everolimus 10 mg QD | Arm B: Single-agent MLN0128 30 mg QW | Arm C: Combination of MLN0128 4 mg QD + MLN1117 200 mg QD
Number analyzed (Participants) | 32 | 32 | 31
Participants | 32 | 30 | 31

3. Secondary Outcome: Overall Survival (OS)
Description: Overall survival in months was defined as the time from the date of randomization to the date of death.
Time Frame: From first dose of study drug through 30 days after the last dose of study drug (up to 51 months)
Population: Full Analysis Set included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Single-agent Everolimus 10 mg QD | Arm B: Single-agent MLN0128 30 mg QW | Arm C: Combination of MLN0128 4 mg QD + MLN1117 200 mg QD
Number analyzed (Participants) | 32 | 32 | 32
months | 22.4 [8.2 to NA] — The upper limit of confidence interval (CI) was not estimable due to fewer number of participants with event. | 16.2 [9.0 to 19.9] | 18.1 [6.2 to 23.4]
Statistical Analysis 1: Comparison: Arm A: Single-agent Everolimus 10 mg QD vs Arm B: Single-agent MLN0128 30 mg QW; Test type: Superiority; p = 0.212, Stratified Log-rank Test; Hazard Ratio (HR) = 1.76, 95% CI 2-sided [0.89 to 3.49] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Arm A: Single-agent Everolimus 10 mg QD vs Arm C: Combination of MLN0128 4 mg QD + MLN1117 200 mg QD; Test type: Superiority; p = 0.546, Stratified Log-rank Test; Hazard Ratio (HR) = 1.51, 95% CI 2-sided [0.77 to 2.98] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Time-to-progression (TTP)
Description: TTP in months is defined as the time from the date of randomization to the date of first documentation of progression. Per RECIST v1.1, PD was defined as at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: From first dose of study drug up to disease progression or death (up to 51 months)
Population: Full Analysis Set included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Single-agent Everolimus 10 mg QD | Arm B: Single-agent MLN0128 30 mg QW | Arm C: Combination of MLN0128 4 mg QD + MLN1117 200 mg QD
Number analyzed (Participants) | 32 | 32 | 32
months | 3.8 [2.0 to 15.6] | 3.5 [1.9 to 7.4] | 3.7 [1.9 to 10.5]
Statistical Analysis 1: Comparison: Arm A: Single-agent Everolimus 10 mg QD vs Arm B: Single-agent MLN0128 30 mg QW; Test type: Superiority; p = 0.156, Log Rank; Hazard Ratio (HR) = 1.57, 95% CI 2-sided [0.81 to 3.05] — HR obtained by stratified Cox proportion hazard model adjusted for prior lines of therapy and the International Metastatic Renal Cell Carcinoma Database Consortium risk category. A hazard ratio < 1 indicates an advantage compared to Everolimus
Statistical Analysis 2: Comparison: Arm A: Single-agent Everolimus 10 mg QD vs Arm C: Combination of MLN0128 4 mg QD + MLN1117 200 mg QD; Test type: Superiority; p = 0.667, Log Rank; Hazard Ratio (HR) = 1.42, 95% CI 2-sided [0.72 to 2.79] — [estimate comment as in outcome 4, analysis 1]

5. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants among response evaluable analysis set who achieve a best overall response of complete response (CR) or partial response (PR) based on investigators assessment of response following RECIST 1.1. CR was defined as disappearance of all target lesions, non-target lesions, no new lesions, and normalization of tumor marker level. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, no progression in non-target lesion, and no new lesions.
Time Frame: From first dose of study drug to disease progression or death (up to 51 months)
Population: Response Evaluable Analysis Set included participants who receive at least 1 dose of study drug, have measurable disease at Baseline and have 1 postbaseline disease assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Arm A: Single-agent Everolimus 10 mg QD | Arm B: Single-agent MLN0128 30 mg QW | Arm C: Combination of MLN0128 4 mg QD + MLN1117 200 mg QD
Number analyzed (Participants) | 32 | 32 | 31
percentage of participants | 15.6 | 0 | 6.5
Statistical Analysis 1: Comparison: Arm A: Single-agent Everolimus 10 mg QD vs Arm C: Combination of MLN0128 4 mg QD + MLN1117 200 mg QD; As prespecified in the protocol, the statistical analysis was performed between arms - Arm A: Single-agent Everolimus 10 mg QD and Arm C: Combination of MLN0128 4 mg QD + MLN1117 200 mg QD only; Test type: Superiority; Odds Ratio (OR) = 0.41, 95% CI 2-sided [0.08 to 2.22] — Odds ratio and 95% CI were obtained using a stratified CMH model with prior lines of therapy and the international metastatic renal cell carcinoma database consortium risk category; As prespecified in protocol, the statistical analysis was performed between arms - Arm A: Single-agent Everolimus 10 mg QD and Arm C: Combination of MLN0128 4 mg QD + MLN1117 200 mg QD only for this outcome measure

6. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: CBR is defined as the percentage of participants who achieve a best response of CR, PR or stable disease (SD) of any duration. CR was defined as disappearance of all target lesions, non-target lesions, no new lesions, and normalization of tumor marker level. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, no progression in non-target lesion, and no new lesions. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
Time Frame: From first dose of study drug up to disease progression or death (up to 51 months)
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Arm A: Single-agent Everolimus 10 mg QD | Arm B: Single-agent MLN0128 30 mg QW | Arm C: Combination of MLN0128 4 mg QD + MLN1117 200 mg QD
Number analyzed (Participants) | 32 | 32 | 31
percentage of participants | 62.5 | 50.0 | 54.8
Statistical Analysis 1: Comparison: Arm A: Single-agent Everolimus 10 mg QD vs Arm B: Single-agent MLN0128 30 mg QW; Test type: Superiority; Odds Ratio (OR) = 0.64, 95% CI 2-sided [0.24 to 1.69] — Odds ratio and 95% CI was obtained using a stratified CMH model with prior lines of therapy and the international metastatic renal cell carcinoma database consortium risk category
Statistical Analysis 2: Comparison: Arm A: Single-agent Everolimus 10 mg QD vs Arm C: Combination of MLN0128 4 mg QD + MLN1117 200 mg QD; Test type: Superiority; Odds Ratio (OR) = 0.79, 95% CI 2-sided [0.28 to 2.21] — [estimate comment as in outcome 6, analysis 1]

7. Secondary Outcome: CBR With SD Duration of at Least 16 Weeks
Description: CBR with SD duration of at least 4 months (CBR-16) was defined as the percentage of participants who achieve CR or PR of any duration or have SD with duration of at least 16 weeks. CR was defined as disappearance of all target lesions, non-target lesions, no new lesions, and normalization of tumor marker level. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, no progression in non-target lesion, and no new lesions. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
Time Frame: Up to Week 16
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Arm A: Single-agent Everolimus 10 mg QD | Arm B: Single-agent MLN0128 30 mg QW | Arm C: Combination of MLN0128 4 mg QD + MLN1117 200 mg QD
Number analyzed (Participants) | 32 | 32 | 31
percentage of participants | 40.6 | 25.0 | 29.0
Statistical Analysis 1: Comparison: Arm A: Single-agent Everolimus 10 mg QD vs Arm B: Single-agent MLN0128 30 mg QW; Test type: Superiority; Odds Ratio (OR) = 0.47, 95% CI 2-sided [0.16 to 1.38] — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Arm A: Single-agent Everolimus 10 mg QD vs Arm C: Combination of MLN0128 4 mg QD + MLN1117 200 mg QD; Test type: Superiority; Odds Ratio (OR) = 0.60, 95% CI 2-sided [0.20 to 1.80] — [estimate comment as in outcome 6, analysis 1]

ADVERSE EVENTS:
Time Frame: All-cause mortality: From first dose of study drug through end of the study (up to 51 months); Serious and other (non-serious) AEs: From first dose of study drug through 30 days after the last dose of study drug (up to 31 months)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. All-cause mortality: Data is reported for Full Analysis Set, defined as all randomized participants (N= 32, 32, 32). Adverse Events: Data for is reported for Safety Analysis Set, including participants who received >=1 dose of study drug.
Arm/Group | Arm A: Single-agent Everolimus 10 mg QD | Arm B: Single-agent MLN0128 30 mg QW | Arm C: Combination of MLN0128 4 mg QD + MLN1117 200 mg QD
All-Cause Mortality (participants affected / at risk) | 16/32 | 18/32 | 19/32
Serious Adverse Events (participants affected / at risk) | 19/32 | 13/32 | 15/31
Other Adverse Events (participants affected / at risk) | 32/32 | 29/32 | 31/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Single-agent Everolimus 10 mg QD (N=32) | Arm B: Single-agent MLN0128 30 mg QW (N=32) | Arm C: Combination of MLN0128 4 mg QD + MLN1117 200 mg QD (N=31)
Pneumonia (Infections and infestations) | 3 | 0 | 0
Sepsis (Infections and infestations) | 2 | 1 | 0
Septic shock (Infections and infestations) | 0 | 1 | 1
Abscess jaw (Infections and infestations) | 1 | 0 | 0
Pulmonary sepsis (Infections and infestations) | 0 | 1 | 0
Asthenia (General disorders) | 0 | 2 | 1
General physical health deterioration (General disorders) | 1 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 1
Fatigue (General disorders) | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 2 | 1
Chronic kidney disease (Renal and urinary disorders) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 2
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 1 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 1
Infarction (Vascular disorders) | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0
Cerebellar haemorrhage (Nervous system disorders) | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Single-agent Everolimus 10 mg QD (N=32) | Arm B: Single-agent MLN0128 30 mg QW (N=32) | Arm C: Combination of MLN0128 4 mg QD + MLN1117 200 mg QD (N=31)
Nausea (Gastrointestinal disorders) | 7 | 22 | 17
Vomiting (Gastrointestinal disorders) | 7 | 14 | 13
Diarrhoea (Gastrointestinal disorders) | 13 | 8 | 11
Constipation (Gastrointestinal disorders) | 9 | 12 | 5
Stomatitis (Gastrointestinal disorders) | 12 | 6 | 3
Abdominal pain (Gastrointestinal disorders) | 5 | 5 | 6
Dyspepsia (Gastrointestinal disorders) | 4 | 4 | 3
Dry mouth (Gastrointestinal disorders) | 1 | 2 | 5
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 1 | 3
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1 | 2
Mouth ulceration (Gastrointestinal disorders) | 3 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 2 | 0
Asthenia (General disorders) | 19 | 12 | 9
Fatigue (General disorders) | 10 | 6 | 12
Pyrexia (General disorders) | 10 | 3 | 5
Chest pain (General disorders) | 2 | 3 | 1
Influenza like illness (General disorders) | 4 | 1 | 1
Chills (General disorders) | 2 | 2 | 1
Oedema peripheral (General disorders) | 4 | 0 | 0
Pain (General disorders) | 1 | 1 | 2
Peripheral swelling (General disorders) | 3 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 15 | 10 | 11
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 4 | 8
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 5 | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 2 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 2 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 1 | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 3 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Iron deficiency (Metabolism and nutrition disorders) | 2 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 12 | 6
Rash (Skin and subcutaneous tissue disorders) | 3 | 3 | 5
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 6 | 2 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 4 | 0 | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 1 | 3
Erythema (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 | 10 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 10 | 3
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Weight decreased (Investigations) | 4 | 9 | 5
Blood creatinine increased (Investigations) | 2 | 3 | 2
Alanine aminotransferase increased (Investigations) | 0 | 1 | 4
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 4
Blood lactate dehydrogenase increased (Investigations) | 1 | 2 | 0
Amylase increased (Investigations) | 2 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 2
Haemoglobin decreased (Investigations) | 2 | 0 | 0
Lipase increased (Investigations) | 2 | 0 | 0
Headache (Nervous system disorders) | 6 | 4 | 4
Dizziness (Nervous system disorders) | 3 | 4 | 0
Dysgeusia (Nervous system disorders) | 3 | 0 | 3
Presyncope (Nervous system disorders) | 3 | 0 | 0
Tremor (Nervous system disorders) | 1 | 0 | 2
Memory impairment (Nervous system disorders) | 2 | 0 | 0
Somnolence (Nervous system disorders) | 2 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 7 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 2 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 1 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Urinary tract infection (Infections and infestations) | 2 | 2 | 2
Influenza (Infections and infestations) | 2 | 0 | 2
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 2
Pneumonia (Infections and infestations) | 2 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 2 | 0
Nasopharyngitis (Infections and infestations) | 2 | 0 | 0
Hypertension (Vascular disorders) | 6 | 3 | 4
Hypotension (Vascular disorders) | 4 | 1 | 1
Anaemia (Blood and lymphatic system disorders) | 4 | 6 | 4
Leukocytosis (Blood and lymphatic system disorders) | 2 | 0 | 0
Anxiety (Psychiatric disorders) | 3 | 2 | 2
Insomnia (Psychiatric disorders) | 3 | 2 | 2
Haematuria (Renal and urinary disorders) | 2 | 1 | 1
Dysuria (Renal and urinary disorders) | 2 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 5 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In general, Investigators may publish clinical data after the earlier of (i) publication by the Sponsor or (ii) 12 months following the abandonment, early termination or database lock; provided a copy of the publication provided to Sponsor at least 30 days ahead of publication, the Sponsor's confidential information is removed as may be requested by Sponsor and Investigator defers publication for up to 60 days in the event Sponsor provides notice that it intends to file a patent application.

DOCUMENTS (2):
  • Study Protocol (2018-12-03): https://cdn.clinicaltrials.gov/large-docs/20/NCT02724020/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-03): https://cdn.clinicaltrials.gov/large-docs/20/NCT02724020/SAP_001.pdf